CLINICAL TRIAL: NCT01003860
Title: Comparison Of 0.5% Vs. 0.75% Ropivacaine Interscalene Brachial Plexus Block (ISB) Prior To Elective Total Shoulder Replacement Surgery On Use of Analgesic Medication During Post-Discharge Week
Brief Title: Postoperative Analgesia After Shoulder Replacement
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Dean Steinberg, M.D., Thomas Jefferson University
Other Study IDs: PCOM2009-01
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Analgesia
Keywords: postoperative analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 0.5% Ropivicaine (150 mg)
- 0.75% Ropivicaine (225 mg)

SUMMARY:
A comparison was made regarding opioid analgesic usage immediately after elective shoulder replacement and for seven days at home between patients randomly given either 0.5% or 0.75% ropivacaine via interscalene block prior to surgery.

It is hypothesized that no significant difference will exist between both groups with respect to pain medication used in the hospital and for a 7-day period at home.

DETAILED DESCRIPTION:
After IRB approval, 46 patients undergoing elective shoulder replacement surgery were recruited at Methodist Hospital (Philadelphia) for this single blind, randomized pilot study. Consented patients spent 48 hours in-house. They were randomly given either 0.5% or 0.75% ropivacaine via interscalene block (ISB) prior to surgery. After the operation, patients were transferred to the post anesthesia care unit (PACU) and placed on a patient controlled analgesia (PCA) morphine pump: basal rate of 0 mg; bolus of 1 mg; lock-out period of 10 min (maximum dose of 6 mg/hr). If the PCA did not provide adequate analgesia, subjects could also receive a bolus of morphine, 2 to 4 mg i.v., every fifteen minutes for several doses p.r.n. In addition, parameters of the PCA could also be modified in order to allow for increased delivery of morphine (e.g., lock-out of 6 min w/max dose of 10 mg/hr) for patient analgesia. PCA morphine therapy was continued after patient was transferred from the PACU to the patient's recovery room. PCA morphine therapy was discontinued the day after surgery and patients were given oral Percocet tablets for pain management. . Thirty-nine patients successfully completed this part of the study. There was no significant difference (p>0.05) between groups in amount of post-operative medications consumed (PCA morphine and oral analgesics) or post-operative pain.

Upon release, patients were given pain and medication diaries to complete for seven successive days. All patients recorded the total amount of Percocet tablets taken at home each day in addition to pain scores (0-10) in the morning, afternoon and evening. Twenty-seven patients successfully completed this part of the study. There was no significant difference (p>0.05)between groups in regard to pain; however, patients in the higher 0.75% group unexpectedly took more tablets (p<0.05).

Conclusion: The 0.5% ISB dose of ropivacaine was found to be equally efficacious as 0.75%; since this lower concentration would also reduce the risk of serious systemic toxicity, it is recommended for ISB prior to elective shoulder replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total shoulder replacement surgery
* 18 years of age or older
* expected length of stay of at least 24 hours
* able to report pain levels
* able to request medications as needed
* American Society of Anesthesiologist (ASA) physical status classification of P1 or P2

Exclusion Criteria:

* liver disease
* kidney disease
* antidepressant therapy (e.g., for clinical depression and/ or chronic pain syndrome)
* ASA physical status classification of P3 or higher
* pregnancy
* allergy to any medications used to treat patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients undergoing shoulder replacement surgery at Methodist Hospital. Ethnicities and ages of patients varied.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Amount of PCA morphine used by pt | for 24 hours following surgery

SECONDARY OUTCOMES:
Amt of analgesic medication used daily at home for 7 days after discharge from hospital | recorded for 7 days at home following discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dean Steinberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Methodist Hospital, Philadelphia, Pennsylvania, United States